CLINICAL TRIAL: NCT07390630
Title: Community Health Worker Implementation of Transdiagnostic Evidence-based Treatment in Spanish
Brief Title: Community Health Worker Implementation of Transdiagnostic Evidence-based Mental Health Intervention for Spanish-speaking Latine Parents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Sinai Urban Health Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0990; K08MD020100 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety; Traumatic Stress
Keywords: community health workers; implementation science; feasibility; parent mental health
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate CETA (Experimental): Participants will participate in up to 14 weekly 1-hour CETA sessions with a community health worker provider
  Interventions: Behavioral: Common Elements Treatment Approach (CETA)
- Delayed CETA (No Intervention): Participants will receive no treatment during a 5-month period while completing symptom measures mirroring those in the active treatment condition. After the delay, participants will be able to receive the treatment.

INTERVENTIONS:
Behavioral: Common Elements Treatment Approach (CETA) — CETA is a transdiagnostic evidence-based treatment (EBT) designed to be implemented in low-resource settings and delivered by lay providers with little to no prior mental health training (i.e., CHWs). CETA consists of 11 modules that address the most common mental health disorders, including depression, anxiety, and post-traumatic stress. Modules are based on common elements of EBT, and include topics of psychoeducation, behavioral activation, relaxation, cognitive restructuring, exposures, safety planning, and substance use reduction. Designed with non-specialists in mind, CETA materials follow a simple, concrete format, with a 1-5 page "manual" section and 1-2 page "steps sheet" for each module that includes goals, example wording, and guidance for in-session use during implementation. CETA has demonstrated effectiveness in RCTs around the world, but has yet to be examined in the US in the context of CHW implementation.
  Other Names: CETA
  Arms: Immediate CETA

SUMMARY:
The goal of this clinical trial is to learn if it is doable for community health workers (CHWs) to deliver a mental health intervention to Spanish-speaking Latine parents experiencing anxiety, depression, and/or traumatic stress. The main questions it aims to answer are (1) Is it doable for CHWs to deliver the mental health intervention and for Latine parents to participate in the intervention, and (2) does the CHW-delivered intervention work in reducing Latine parents' mental health symptoms.

Researchers will compare Latine parents receiving the intervention to Latine parents not receiving the intervention to see if the CHW-delivered intervention works to improve mental health symptoms.

Participants will:

* Participate in up to 14 weekly 1-hour sessions of the mental health intervention delivered by a CHW. They will be randomized to receive the intervention immediately or after a 5-month delay.
* Participants will complete questionnaires about their symptoms, family and child functioning, as well as about how doable, acceptable, and appropriate they found the intervention
* Participants will also complete a recorded interview about their experience in the intervention

ELIGIBILITY:
INCLUSION criteria for PATIENT participants are:

* 18 years or older
* Identifies as Latine
* Is a caregiver to a child 18 years or younger old living in the same household
* Preference for Spanish services
* Symptom scores in the moderate range for depression, anxiety, and/or PTSD (based on Computerized Adaptive Tests for Mental Health (CAT-MH))

EXCLUSION criteria for PATIENT participants:

* Presence of mania symptoms in the mild range or higher (based on CAT-MH responses)
* Presence of psychosis symptoms in mild range or higher (based on CAT-MH responses)
* Active suicidal ideation (based on CAT-MH responses)
* Depression, anxiety, or PTSD symptoms in the severe range (based on CAT-MH responses)
* Currently receiving psychotherapy services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2027-02 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Patient engagement | Through study completion; over the course of approximately up to 5 months of participant participation
  Number of intervention sessions completed per patient
Fidelity | Completed after each CETA session through study completion, over the course of approximately up to 5 months of participant participation
  CETA Fidelity Monitory System: Session information is documented by the CETA provider, who is trained to document what they did in each session relating to specific steps outlined in each CETA element. Each element in the CETA manual is executed through detailed "steps". Fidelity includes what CETA elements are chosen, when they are delivered, steps completed within each element, and the frequency in which each element is delivered.
Patient intervention retention | Through study completion; over the course of approximately up to 5 months of participant participation
  Number of patients who begin the intervention and go on to complete the intervention
Patient control retention | Through study completion; over the course of approximately up to 5 months of participant participation
  Number of participants assigned to the control condition who remain enrolled at the end of the 5-month delay period
Patient assessment completion | Through study completion; over the course of approximately up to 5 months of participant participation
  Proportion of planned assessments that are completed by patients
Patient intervention feasibility, acceptability, & appropriateness | Patients will complete the mhIST immediately after their last intervention session
  The Mental Health Implementation Science Tools (mhIST), consumer version measures domains of acceptability, appropriateness, and feasibility via self-report by those receiving an intervention. The mhIST uses a four-point Likert scale with the options of "Not at all," "A little bit," "A moderate amount," and "A lot."
Provider intervention feasibility, acceptability, & appropriateness | After approximately 2 years of intervention delivery
  The Mental Health Implementation Science Tools (mhIST), provider version measures domains of acceptability, appropriateness, and feasibility via self-report by those delivering an intervention. The mhIST uses a four-point Likert scale with the options of "Not at all," "A little bit," "A moderate amount," and "A lot."

SECONDARY OUTCOMES:
Patient mental health symptoms: Baseline | Baseline pre-randomization
  Computerized Adaptive Testing (CAT) for Mental Health (CAT-MH): The CAT-MH is a suite of multidimensional item response theory (IRT) based CATs for the dimensional measurement of symptoms of depression, anxiety, and PTSD, amongst others. The CAT-MH generates a score and accompanying severity band for each disorder module based on patient report.
Patient mental health symptoms: Monthly | Completed monthly while receiving the intervention or during the 5-month delay period (depending on randomization assignment)
  Computerized Adaptive Testing (CAT) for Mental Health (CAT-MH): The CAT-MH is a suite of multidimensional item response theory (IRT) based CATs for the dimensional measurement of symptoms of depression, anxiety, and PTSD, amongst others. The CAT-MH generates a score and accompanying severity band for each disorder module based on patient report.
Patient mental health symptoms: Post-intervention | Completed immediately after the last intervention session
  Computerized Adaptive Testing (CAT) for Mental Health (CAT-MH): The CAT-MH is a suite of multidimensional item response theory (IRT) based CATs for the dimensional measurement of symptoms of depression, anxiety, and PTSD, amongst others. The CAT-MH generates a score and accompanying severity band for each disorder module based on patient report.
Patient mental health symptoms: 1-month post-intervention | Completed 1 month after the last intervention session
  Computerized Adaptive Testing (CAT) for Mental Health (CAT-MH): The CAT-MH is a suite of multidimensional item response theory (IRT) based CATs for the dimensional measurement of symptoms of depression, anxiety, and PTSD, amongst others. The CAT-MH generates a score and accompanying severity band for each disorder module based on patient report.
Patient mental health symptoms: 3-months post-intervention | Completed 3 months after the last intervention session
  Computerized Adaptive Testing (CAT) for Mental Health (CAT-MH): The CAT-MH is a suite of multidimensional item response theory (IRT) based CATs for the dimensional measurement of symptoms of depression, anxiety, and PTSD, amongst others. The CAT-MH generates a score and accompanying severity band for each disorder module based on patient report.
Patient quality of life: Baseline | Baseline pre-randomization
  World Health Organization Quality of Life - Abbreviated version (WHOQOL-BREF): patient-report of quality of life across domains of physical health, psychological health, social relationships, and environment, using a 5-point likert scale.
Patient quality of life: Post-intervention | Completed immediately post-intervention
  World Health Organization Quality of Life - Abbreviated version (WHOQOL-BREF): patient-report of quality of life across domains of physical health, psychological health, social relationships, and environment, using a 5-point likert scale.
Patient quality of life: 1-month post-intervention | Completed 1 month post-intervention
  World Health Organization Quality of Life - Abbreviated version (WHOQOL-BREF): patient-report of quality of life across domains of physical health, psychological health, social relationships, and environment, using a 5-point likert scale.
Patient quality of life: 3-month post-intervention | Completed 3 month post-intervention
  World Health Organization Quality of Life - Abbreviated version (WHOQOL-BREF): patient-report of quality of life across domains of physical health, psychological health, social relationships, and environment, using a 5-point likert scale.
Parenting stress: Baseline | Baseline pre-randomization
  Parental Stress Scale (PSS): patient-report of parenting stress across three scales -- parental distress, parent-child dysfunctional interaction, and difficult child -- using a 1 (strongly disagree) - 5 (strongly agree) likert scale
Parenting stress: Post-intervention | Completed immediately after the last intervention session
  Parental Stress Scale (PSS): patient-report of parenting stress across three scales -- parental distress, parent-child dysfunctional interaction, and difficult child -- using a 1 (strongly disagree) - 5 (strongly agree) likert scale
Parenting stress: 1-month post-intervention | Completed 1 month after the last intervention session
  Parental Stress Scale (PSS): patient-report of parenting stress across three scales -- parental distress, parent-child dysfunctional interaction, and difficult child -- using a 1 (strongly disagree) - 5 (strongly agree) likert scale
Parenting stress: 3-month post-intervention | Completed 3 months after the last intervention session
  Parental Stress Scale (PSS): patient-report of parenting stress across three scales -- parental distress, parent-child dysfunctional interaction, and difficult child -- using a 1 (strongly disagree) - 5 (strongly agree) likert scale
Child mental health: Baseline | Baseline pre-randomization
  Strengths and Difficulties Questionnaire (SDQ): Patient-report of child's behavioral functioning across five scales (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships; and prosocial behaviors) for each of their children using a 3-point likert scale (not true, somewhat true, & certainly true).
Child mental health: Post-intervention | Completed immediately after the last intervention session
  Strengths and Difficulties Questionnaire (SDQ): Patient-report of child's behavioral functioning across five scales (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships; and prosocial behaviors) for each of their children using a 3-point likert scale (not true, somewhat true, & certainly true).
Child mental health: 1-month post-intervention | Completed 1 month after the last intervention session
  Strengths and Difficulties Questionnaire (SDQ): Patient-report of child's behavioral functioning across five scales (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships; and prosocial behaviors) for each of their children using a 3-point likert scale (not true, somewhat true, & certainly true).
Child mental health: 3-month post-intervention | Completed 3 months after the last intervention session
  Strengths and Difficulties Questionnaire (SDQ): Patient-report of child's behavioral functioning across five scales (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships; and prosocial behaviors) for each of their children using a 3-point likert scale (not true, somewhat true, & certainly true).
Family functioning: Baseline | Baseline pre-randomization
  Family Relations Scale: participant-report of family functioning across three scales -- family cohesion, support, and organization -- using a 4-point likert scale (1: not true at all - 4: almost always or always true)
Family functioning: Post-intervention | Completed immediately after the last intervention session
  Family Relations Scale: patient-report of family functioning across three scales -- family cohesion, support, and organization -- using a 4-point likert scale (1: not true at all - 4: almost always or always true)
Family functioning: 1-month post-intervention | Completed 1 month after the last intervention session
  Family Relations Scale: patient-report of family functioning across three scales -- family cohesion, support, and organization -- using a 4-point likert scale (1: not true at all - 4: almost always or always true)
Family functioning: 3-month post-intervention | Completed 3 months after the last intervention session
  Family Relations Scale: patient-report of family functioning across three scales -- family cohesion, support, and organization -- using a 4-point likert scale (1: not true at all - 4: almost always or always true)

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets containing quantitative questionnaire data from patient participants will be made available via an open institutional repository. Specific de-identified data elements will include demographic, administrative (condition assignment, attendance, fidelity), clinical (symptom questionnaires about mental health, well being, family, and child functioning), and implementation (intervention acceptability, feasibility) data.
Supporting Information: Study Protocol
Time Frame: April 2029 to March 2034
Access Criteria: Data will be uploaded to an institutional repository that is open to the general public.